CLINICAL TRIAL: NCT04129814
Title: The Effects of Non -Surgical Periodontal Treatment on The Severity of Erectile Dysfunction (Randomized Controlled Clinical Trial)
Brief Title: The Effects of Non -Surgical Periodontal Treatment on The Severity of Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taibah University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Yasser El Makaky, Associated professor, Taibah University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: periodontal therapy and IIEF
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Periodontitis; Erectile Dysfunction
Keywords: Chronic periodontitis; Prognosis; Erectile Dysfunction
MeSH Terms: conditions — Periodontitis; Erectile Dysfunction; Chronic Periodontitis

STUDY DESIGN:
Intervention Model Description: After periodontal and medical screening, all eligible patients will informed of potential risks, study objective, and benefits of their participation in this study. Non-surgical periodontal treatment consisted of oral hygiene instructions (OHI), single session full-mouth scaling and root planing (SRP) that will be performed by the same periodontist using Gracey curettes (Hu-Friedy, Chicago, IL, USA) and ultrasonic apparatus (Cavitron Select SPC, Dentsply professional, New York, USA) for all participants within a test group at baseline and after three months for patients in a control group because of ethical reasons. Therefore, no periodontal treatment will be performed during the follow-up period in control group.
Who Masked: Participant
Masking Description: Statistical software (STATA 13.1, Stata Corp, Texas, USA) was used for random and equal stratification of the participants according to their mean values of IIEF, and this identify to which group the patients were enrolled, using 1:1 allocation ratio.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): Non-surgical periodontal treatment consisted of oral hygiene instructions (OHI), single session full-mouth scaling and root planing (SRP)
  Interventions: Procedure: Non surgical periodontal therapy
- control group (No Intervention): no periodontal treatment was performed during the follow-up period in the control group.

INTERVENTIONS:
Procedure: Non surgical periodontal therapy — single session full-mouth scaling and root planing
  Arms: test group

SUMMARY:
The aim of the present study is to study the influence of periodontal therapy (non-surgical) on the severity of erectile dysfunction(ED) among patients with chronic periodontitis and moderate or severe ED.

DETAILED DESCRIPTION:
there no sufficient data to determine a possible link between erectile dysfunction ( ED) and periodontitis. Therefore, the purpose of this clinical trial is to study the influence of periodontal therapy (non-surgical) on the severity of ED among patients with chronic periodontitis and moderate or severe ED.

Sample size: The total number of patients in the current trial will be 140 to requite dropout rate during follow-up period.

Patients and study design:

The current trial is a single-blinded, randomized, parallel, controlled clinical study.

The patients with severe or moderate ED will selected from attendants of Andrology Outpatients Clinic, Tanta University Hospital and will referred to Periodontology Department, Tanta University. Statistical software (STATA 13.1, Stata Corp, Texas, USA) will be used on study participants for random allocation that identify to which group the patients will enrolled, using 1:1 allocation ratio.

Intervention protocol The patients will included in this study if they met the inclusion criteria. The IIEF is an appropriate questionnaire that is used for assessment of men sexual function, especially the ED. . Subjects with scores > 25 will assessed as men with normal sexual function while those with scores ≤ 25 will diagnosed as patients with ED. Following this, participants will directed to periodontology department to assess their periodontal health . After periodontal screening, all eligible patients will informed of potential risks, study objective, and benefits of their participation in this study. Non-surgical periodontal treatment that will be performed by the same periodontist for all participants within a test group at baseline and after three months for patients in a control group. Therefore, no periodontal treatment will be performed during the follow-up period in control group. D

Clinical and periodontal evaluation Thorough medical history, data on age, gender and socio-demographic characteristics will be gathered for all participants in studied groups at baseline. A full-mouth periodontal screening will be carried out by one specialist using a manual probe (Hu-Friedy, Chicago, IL, USA). Prior the current study, test-retest exercises will be performed in 20 patients to assess intra-examiner calibration. The periodontal parameters will be assessed at baseline and at 3 months that consist of PD, CAL, visible dental plaque (will be assessed at 4 sites per each tooth using a probe and will be recorded as present or absent) and bleeding on probing (BOP) (will be recorded as ratio of sites displaying bleeding after light probing) 10. After exclusion of third molars; for each tooth BOP, CAL and PD will be monitored at 6 sites. The IIEF scores will be recorded at baseline and 3 months for both groups.

Cytokine collection and evaluation:

Quantitative assessment of TNF-α in saliva and serum will be done by commercially available kit (Ray Bio Human TNF-α Enzyme Immunoassay).

ELIGIBILITY:
Inclusion Criteria:

* Age from 30 to 40 years
* Diagnosis with chronic periodontitis using the classification system of (Armitage, 1999)19 for periodontal diseases
* Presence of at least sixth permanent teeth excluding the third molars20
* Clinical attachment level (CAL) and pocket depth (PD) ≥4 mm in more than 30% of sites19
* Severe or moderate ED
* Male patients
* Married

Exclusion Criteria:

* Alcoholism and smokers
* Presence of any systemic disorders that may affect ED or periodontal health such as heart disease, diabetes mellitus, and hypertension18
* Antimicrobial therapies in the last 6 months
* Periodontal treatment in the last 6 months
* Drug therapy that may cause ED as side effects such as atenolol and hydrochlorothiazide

Ages: 30 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
changes in the severity of Erectile Dysfunction | 3 months
  changes in the severity of Erectile Dysfunction diagnosed by International Index of Erectile Dysfunction between test and control groups. Subjects with scores > 25 were assessed as men with normal sexual function while those with scores ≤ 25 were diagnosed as patients with erectile dysfunction.severe with a score from 6 to 10, moderate (11-16) and mild (17-25)

SECONDARY OUTCOMES:
changes in mean values of TNF-α in serum.Quantitative assessment of TNF-α in serum was done by a commercially available kit (Ray Bio Human TNF-α Enzyme Immunoassay),and was expressed as pg/mL. | 3 months
  changes between groups throughout the follow-up period in mean values of TNF-α level in serum .
changes in mean values of TNF-α in saliva | 3 momths
  changes between groups throughout the follow-up period in mean values of TNF-α level in saliva .Quantitative assessment of TNF-α in saliva and serum was done by a commercially available kit (Ray Bio Human TNF-α Enzyme Immunoassay). and was expressed as pg/mL.
changes in mean values of Clinical attachment level | 3 months
  changes between groups throughout the follow-up period in mean values of Clinical attachment level (distance from the base of the pocket to cement-enamel junction) which measured in milmiters using a manual probe (Hu-Friedy, Chicago, IL, USA).